CLINICAL TRIAL: NCT06921304
Title: BASE-DIET: a Randomized Clinical Trial to Examine the Impact of a Dietary-nutritional Intervention on Body Weight Recovery, Metabolic Parameters, and Body Composition in Patients With a New Diagnosis of Graves' Disease
Brief Title: BASE-DIET: a Study on Nutritional Intervention in Patients With Graves' Disease
Acronym: BASEDIET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Laura Croce, Professor, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BASE-DIET 01
Record Dates: First submitted 2025-04-01; First posted 2025-04-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Graves Disease
Keywords: graves disease; diet; body weight; PREDIMED
MeSH Terms: conditions — Graves Disease; Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Medical Care (UMC) (No Intervention): Usual Medical Care for Graves' Disease and general lifestyle advice
- Intensive Lifestyle Intervention (ILI) (Experimental): Usual Medical Care for Graves' Disease plus a personalized diet and lifestyle counseling
  Interventions: Behavioral: Intensive Lifestyle Intervention

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — ILI combines a low-calorie dietary approach with improved lifestyle and physical activity, in addition to usual medical care. Behavioral support for lifestyle intervention will also be provided.
  Arms: Intensive Lifestyle Intervention (ILI)

SUMMARY:
The goal of this clinical trial is to determine whether a structured dietary-nutritional intervention can prevent excessive weight regain and improve body composition and lifestyle habits in adults recently diagnosed with Graves' disease (Basedow's disease).

The main questions it aims to answer are:

* Can a dietary intervention prevent patients from regaining more than 1 kg above their pre-disease body weight after restoring euthyroidism?
* Does the intervention lead to improvements in body composition, dietary habits, and adherence to the Mediterranean diet? Researchers will compare patients receiving an Intensive Lifestyle Intervention (ILI) including a personalized diet and lifestyle counseling to patients receiving Usual Medical Care (UMC) with general lifestyle advice to see if the dietary intervention results in less weight regain and better metabolic and anthropometric outcomes.

Participants will:

* Receive antithyroid medication as standard medical care.
* Be randomized into either the intervention group (ILI) or control group (UMC).

If in the ILI group, participants will:

* Receive an individual nutritional consultation within 1 week of enrollment.
* Follow a personalized Mediterranean-style low-energy diet.
* Attend follow-up visits at 3, 6, 9, and 12 months for:

  * Dietary adherence and lifestyle assessments.
  * Anthropometric measurements (weight, BMI, waist/hip circumference).
  * Bioimpedance analysis (at 6 and 12 months) for body composition.
  * Dietary intake logs and adherence assessments (3-day food diary).

If in the UMC group, participants will:

* Receive routine clinical management for Graves' disease.
* Complete basic dietary and lifestyle questionnaires at baseline and 12 months.
* Undergo anthropometric measurements and bioimpedance at T0 and at the end of study.

This study aims to provide evidence on the role of nutritional support in managing weight and metabolic risks in patients undergoing treatment for Graves' disease.

DETAILED DESCRIPTION:
What is the BASE-DIET Study? The BASE-DIET study is a clinical trial looking at how a healthy diet and lifestyle program can help people newly diagnosed with Graves' disease (an autoimmune thyroid condition) manage weight changes and improve their health during and after treatment.

Graves' disease often causes weight loss when it's active. But after treatment, many people gain back the weight-and sometimes even more than they had before. This study wants to find out if a personalized diet and lifestyle approach can help prevent that excessive weight gain and promote better health outcomes.

Why is this study important? When thyroid function is brought back to normal (called "euthyroidism"), many patients regain weight. In fact, up to 80% of patients report weight gain after treatment, which can impact self-esteem and health.

Some research shows this weight gain might go beyond what people weighed before getting sick. This study wants to see whether a structured diet and lifestyle program can make a positive difference compared to the usual medical care alone.

Who is participating in the study?

Adults newly diagnosed with Graves' disease at endocrinology clinics in Italy are invited to take part. Participants must:

* Be over 18 years old
* Have been diagnosed within the previous month
* Have a BMI between 16 and 35
* Be willing to commit to a 1-year program They cannot participate if they are pregnant, have certain health conditions, or are already taking weight-related medications.

How is the study organized?

The study randomly assigns people to one of two groups:

1. Intervention Group (ILI) - This group receives:

   * Personalized nutrition counseling by a licensed dietitian
   * A Mediterranean-style, low-calorie diet plan
   * Support on physical activity and lifestyle
   * Follow-up appointments at 3, 6, 9, and 12 months
2. Control Group (UMC) - This group receives:

   * Standard medical care for Graves' disease
   * General lifestyle and diet tips (no personalized plan)
   * Two check-ins at the beginning and end of the 12-month period What is being measured? The main goal (primary outcome) is to see if people in the intervention group are less likely to gain more than 1 kg over their pre-disease weight after 12 months.

Secondary goals include:

* Changes in Body Mass Index (BMI)
* Body composition (muscle vs. fat mass)
* Waist-to-hip ratio
* Adherence to a Mediterranean diet
* Improved eating habits and quality of life What happens during follow-up?

At each check-up, researchers will:

* Measure weight, height, waist and hip size
* Use a body composition test (bioimpedance analysis)
* Review a 3-day food diary
* Ask about physical activity and lifestyle changes
* Check how closely participants follow the prescribed diet Only the intervention group receives repeated, in-depth dietary coaching. How long does the study last? The full study duration for each participant is 12 months, with an extended follow-up period for data collection.

How many people are in the study? The study plans to enroll 60 people (30 in each group), which accounts for a small number of possible dropouts.

Is the study safe and ethical?

Yes. It follows strict ethical guidelines:

* All participants give written informed consent
* Privacy is fully protected
* Participation is voluntary, and people can leave at any time There are no outside sponsors-it's a non-profit, academic study led by IRCCS Maugeri in Pavia, Italy.

What will happen with the results?

Results will be:

* Published in scientific journals
* Shared at medical conferences
* Made available to the public The goal is to better understand how diet can help people with Graves' disease manage their weight and improve their recovery.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Graves' disease in an endocrinology setting based on the presence of thyrotoxicosis and positive TRAb antibodies.
* Diagnosis of Graves' disease within 1 month prior to randomization.
* BMI > 16 kg/m² and < 35 kg/m² at the time of the first visit for Graves' disease.
* Age > 18 years.
* Ability to commit to the duration of the study.
* Ability to provide informed consent and willingness to participate in the study.

Exclusion Criteria

* Relapse of Graves' disease or thyrotoxicosis not related to Graves' disease.
* Any serious cardiovascular or renal event in the last 6 months.
* Current pregnancy, breastfeeding, or planning pregnancy during the study period.
* Any condition potentially leading to fluid overload such as heart failure (NYHA class > I) or liver cirrhosis.
* Previously diagnosed significant psychiatric disorder (e.g., schizophrenia, post-traumatic stress disorder, obsessive-compulsive disorder).
* Active eating disorder.
* Uncontrolled depression.
* Uncontrolled epilepsy.
* Known cause of malabsorption (including uncontrolled celiac disease, lactose intolerance, or inflammatory bowel disease).
* Ongoing therapy with weight-modifying medications (e.g., GLP-1 analogs, metformin).
* Estimated BMI before disease onset < 18 kg/m². This parameter will be calculated based on the "estimated pre-disease body weight" as reported by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Body weight increase vs pre-disease weight | Through study completion, an average of 1 year
  Weight gain compared to the estimated pre-disease body weight. A 'failure' will be defined as a weight gain of more than 1 kg above the patient-reported estimated pre-disease body weight, assessed 12 months after the start of the study. Body weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
BMI changes | Through study completion, an average of 1 year
  Direct comparison of the BMI achieved at the end of the study period between the two groups, with subsequent calculation of weight gain relative to baseline weight. Weight change will be assessed as the difference between the weight measured in kilograms at the end of the study and that measured at the beginning, expressed as a percentage of the initial weight. Body weight and height will be combined to report BMI in kg/m^2
Adherence to the Mediterranean Diet | Through study completion, an average of 1 year
  A successful outcome will be defined as an improvement in adherence scores based on the PREDIMED questionnaire.
Changes in body composition parameters | Through study completion, an average of 1 year
  This will be defined as the normalization of abnormal values of fat mass percentage, lean mass, or total body water detected at baseline (T0). For participants with optimal values at T0, success will be defined as maintaining optimal parameters; worsening of these parameters will be considered a failure.
Changes in waist-to-hip ratio | Through study completion, an average of 1 year
  A successful outcome will be defined as an improvement in waist-to-hip ratio in participants with abnormal values at baseline. For those with optimal values at T0, maintaining optimal parameters will be considered a success, while deterioration will be considered a failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Maugeri IRCCS, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Croce L, Pallavicini C, Busca N, Cali B, Bellastella G, Coperchini F, Magri F, Chiovato L, Cena H, Rotondi M. Pre-surgery dietician counseling can prevent post-thyroidectomy body weight gain: results of an intervention trial. Endocrine. 2023 Aug;81(2):246-251. doi: 10.1007/s12020-023-03365-z. Epub 2023 Apr 19. PMID 37074559
- [Background] Pijl H, de Meijer PH, Langius J, Coenegracht CI, van den Berk AH, Chandie Shaw PK, Boom H, Schoemaker RC, Cohen AF, Burggraaf J, Meinders AE. Food choice in hyperthyroidism: potential influence of the autonomic nervous system and brain serotonin precursor availability. J Clin Endocrinol Metab. 2001 Dec;86(12):5848-53. doi: 10.1210/jcem.86.12.8112. PMID 11739450
- [Background] van Veenendaal NR, Rivkees SA. Treatment of pediatric Graves' disease is associated with excessive weight gain. J Clin Endocrinol Metab. 2011 Oct;96(10):3257-63. doi: 10.1210/jc.2011-1601. Epub 2011 Aug 17. PMID 21849528
- [Background] Chng CL, Lim AY, Tan HC, Kovalik JP, Tham KW, Bee YM, Lim W, Acharyya S, Lai OF, Chong MF, Yen PM. Physiological and Metabolic Changes During the Transition from Hyperthyroidism to Euthyroidism in Graves' Disease. Thyroid. 2016 Oct;26(10):1422-1430. doi: 10.1089/thy.2015.0602. Epub 2016 Sep 7. PMID 27465032
- [Background] Kim MJ, Cho SW, Choi S, Ju DL, Park DJ, Park YJ. Changes in Body Compositions and Basal Metabolic Rates during Treatment of Graves' Disease. Int J Endocrinol. 2018 May 3;2018:9863050. doi: 10.1155/2018/9863050. eCollection 2018. PMID 29853888
- [Background] Krassas GE, Pontikides N, Loustis K, Koliakos G, Constantinidis T, Panidis D. Resistin levels in hyperthyroid patients before and after restoration of thyroid function: relationship with body weight and body composition. Eur J Endocrinol. 2005 Aug;153(2):217-21. doi: 10.1530/eje.1.01963. PMID 16061827
- [Background] Hoogwerf BJ, Nuttall FQ. Long-term weight regulation in treated hyperthyroid and hypothyroid subjects. Am J Med. 1984 Jun;76(6):963-70. doi: 10.1016/0002-9343(84)90842-8. PMID 6731468
- [Background] Alton S, O'Malley BP. Dietary intake in thyrotoxicosis before and after adequate carbimazole therapy; the impact of dietary advice. Clin Endocrinol (Oxf). 1985 Nov;23(5):517-20. doi: 10.1111/j.1365-2265.1985.tb01111.x. PMID 4085132
- [Background] Lonn L, Stenlof K, Ottosson M, Lindroos AK, Nystrom E, Sjostrom L. Body weight and body composition changes after treatment of hyperthyroidism. J Clin Endocrinol Metab. 1998 Dec;83(12):4269-73. doi: 10.1210/jcem.83.12.5338. PMID 9851762